CLINICAL TRIAL: NCT05207345
Title: Effectiveness of Core Stability Training on Trunk Control in Patients With Post-hemorrhagic Stroke
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Marco Monticone, Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG/2021/17872
Record Dates: First submitted 2022-01-11; First posted 2022-01-26 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Hemorrhagic Stroke
Keywords: Hemorrhagic Stroke, Trunk Impairment, Core Stability
MeSH Terms: conditions — Hemorrhagic Stroke

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 90-minute session divided into:
  * 45 minutes of "core stability" treatment
  * 45 minutes of general rehabilitation (active / active, assisted / passive mobilization, stretching, posture maintenance, postural and autonomy training, cycle ergometer, exercise bike and ambulatory training).
  Interventions: Other: Interventional programme
- General Group (Active Comparator): 90 minutes of general rehabilitation (active / active assisted / passive mobilization, stretching, posture maintenance, postural and autonomy training, cycle ergometer, exercise bike and ambulatory training).
  Interventions: Other: General exercise programme

INTERVENTIONS:
Other: Interventional programme — 90-minute session divided into:
  * 45 minutes of "core stability" treatment
  * 45 minutes of general rehabilitation (active / active, assisted / passive mobilization, stretching, posture maintenance, postural and autonomy training, cycle ergometer, exercise bike and ambulatory training).
  Arms: Experimental Group
Other: General exercise programme — 90 minutes of general rehabilitation (active / active assisted / passive mobilization, stretching, posture maintenance, postural and autonomy training, cycle ergometer, exercise bike and ambulatory training).
  Arms: General Group

SUMMARY:
Stroke is responsible for about 7% of disabilities in the European population. Intracerebral hemorrhage (ICH) represents 15% of stroke cases in Europe. In order to avoid disabling sequelae, an essential role is played by early rehabilitation, which has also proved effective for ICH.

In addition to its role in physical recovery, it plays a fundamental role in the psychological well-being of patients with ICH.

Impairments in trunk function are a common sequela and are related to reduced mobility, balance and functional independence.

Trunk exercises could improve trunk control, postural control, and functional recovery.

The hypothesis is that a specific exercise program, based on core stability, will induce clinically significant and long-term improvements from the point of view of trunk control, and secondly in postural control, disability and quality of life in subjects with hemorrhagic stroke outcomes, versus general physiotherapy, and that these improvements will be maintained at least one year after the intervention.

DETAILED DESCRIPTION:
Stroke is responsible for about 7% of disabilities in the European population, and in particular intracerebral hemorrhage (ICH), whose mortality is higher than ischemic stroke, represents 15% of stroke cases in Europe.

In order to avoid disabling sequelae, an essential role is played by early rehabilitation, which has also proved effective for ICH.

Patients undergoing early rehabilitation within neurorehabilitation units achieve better clinical-functional outcomes than those who receive general medical care; furthermore, in addition to its role in physical recovery, it plays a fundamental role in the psychological well-being of patients with ICH, as these patients tend to be less depressed and anxious than those undergoing standard care.

However, even after intensive rehabilitation functional deficits still exist, making stroke the leading cause of disability in adults globally.

Impairments in trunk function, in particular, are a common sequelae and are related to reduced mobility, balance and functional independence. Therefore, impairments in trunk function can lead to limitations of activity and participation, as well as to increase the risk of falling resulting in further disability, hospitalization and mortality.

The dysfunction of the core, which would significantly affect the function of the trunk, would seem to be linked to a reduction in muscle strength, to a delayed/asymmetrical activation of the muscles, as well as to proprioceptive alterations.

Following this line, trunk exercises could then improve trunk control, postural control, and functional recovery.

Looking at the literature, it has been seen how several randomized controlled trials have focused on the efficacy of trunk training in stroke populations with positive and encouraging results regarding the outcomes achieved within the experimental groups. However, these studies, in addition to including patients with both ischemic and haemorrhagic stroke, did not always equalize the amount of exercise provided with a control group, showing heterogeneity in the exercises administered, and did not consider whether the therapeutic efficacy observed at the end of the treatment is still maintained over the long term.

The hypothesis is that a specific exercise program, based on core stability, will induce clinically significant and long-term improvements from the point of view of trunk control, and secondly in postural control, disability and quality of life in subjects with hemorrhagic stroke outcomes, versus general physiotherapy, and that these improvements will be maintained at least one year after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* haemorrhagic stroke < 3 months, first event
* adulthood (40-75 years)
* ability to maintain the sitting position
* good knowledge of the Italian language

Exclusion Criteria:

* cognitive impairment
* Ashworth score> 2
* Neurodegenerative and/or neuromuscular disorders
* Severe cardiovascular and respiratory instability, systemic diseases

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Trunk Impairment Scale at 8 weeks and 12 months | Questionnaires will be administered before treatment, eight weeks after (post-treatment) and 12 months after the end of treatment (follow-up)
  The Trunk Impairment Scale (TIS) is a 17-item scale that aims to assess the static, dynamic balance and coordination of the trunk. Each item is given a variable score from 0 to 3 in relation to the performance analyzed. The final score can range from a minimum of 0 points to a maximum of 23. The higher the score, the more independent the patient is in performing trunk control. Investigators used the Italian version which proved to be reliable and valid

SECONDARY OUTCOMES:
Change from Baseline Functional Independence Measure (FIM) at 8 weeks and 12 months | Questionnaires will be administered before treatment, eight weeks after (post-treatment) and 12 months after the end of treatment (follow-up)
  FIM describes 18 Activities of daily living (ADLs) associated with motor, cognitive, and sphincteral problems and ranges from 18 (maximal limitation) to 126 (no limitation).
  Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item.
Change from Baseline Berg Balance Scale (BBS) at 8 weeks and 12 months | Questionnaires will be administered before treatment, eight weeks after (post-treatment) and 12 months after the end of treatment (follow-up)
  It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function Final score ranges from 0 (high risk of falling) to 56 (no risk of falling).
Change from Baseline Short-Form Health Survey Questionnaire at 8 weeks and 12 months | Questionnaires will be administered before treatment, eight weeks after (post-treatment) and 12 months after the end of treatment (follow-up)
  Quality of life is assessed using the Italian version of the self-report Short-Form Health Survey with its eight domain scores ranging from 0 (the worst perceived quality of life) to 100 (the best perceived quality of life).
Global Perceived Effect | eight weeks after starting treatment (post-treatment)
  Global Perceived Effect is a self-administered measure of treatment satisfaction consisting of a five-level Likert scale (1=helped a lot, 2=helped, 3=helped only a little, 4=did not help, 5=made things worse).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Monticone, MD, PhD, Study Chair — University of Cagliari
Locations (1):
- University of Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No